CLINICAL TRIAL: NCT04298346
Title: GENIMOC : Neurological Fate, Prematurity and Genetic Susceptibility Factors
Brief Title: Neurological Fate, Prematurity and Genetic Susceptibility Factors
Acronym: GENIMOC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0035
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2021-09

CONDITIONS: Polymorphism, Restriction Fragment Length; Premature; Infertility of Cervical Origin
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
  Interventions: Other: no intervention
- Control
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study could help identify aggravating or protective genetic polymorphisms associated with cerebral palsy. Populations of premature babies at different risk of cerebral palsy could thus be individualized with an impact on their monitoring and on the pathophysiological understanding of the processes leading to neurological lesions.

ELIGIBILITY:
Inclusion Criteria:

* children born prematurely at term <34 weeks between 2008 and 2015
* assessed at the age of 2 within the Growing Together Network in Pays de Loire
* parental consent for the collection of data from their child and for intraoral sampling for the search for genetic factors.

Exclusion Criteria:

* children who died after the age of 2
* children who refused and / or whose parents refused to participate in the study

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children born prematurely at term <34 weeks between 2008 and 2015, and presenting with cerebral palsy at the age of 2 years within the Growing Together Network in Pays de Loire.
  Matching by a propensity score to a population of control children with a comparable probability of developing cerebral palsy but whose examination at 2 years is optimal
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Identify a polymorphism associated with the risk of developing cerebral palsy at 2 years in a regional population of premature infants of gestational age <34 weeks gestation. | 2 years
  frequency of variants within the case and control groups using the statistical criterion "level of significance" (also called p-value and known by the English word "p-value") of 5.10-8

SECONDARY OUTCOMES:
Identify a specific polymorphism of certain forms of cerebral palsy | 2 years
  neurological examination
Develop a prognosis algorithm for the occurrence of cerebral palsy for personalized monitoring in a population at risk. | 2 years
  neurological examination

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided